CLINICAL TRIAL: NCT06096636
Title: National Survey of Young Adult Nutrition
Acronym: NAYAN
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Other Study IDs: GFHNRC340
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Overweight or Obesity
Keywords: Healthy Weight
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participants: Participants will complete survey and dietary assessment.
  Interventions: Other: Study participants

INTERVENTIONS:
Other: Study participants — Participants will complete study survey and dietary assessment.

SUMMARY:
The purpose of this research is to better understand how people's background, habits, and other factors influence their diets and health.

DETAILED DESCRIPTION:
The purpose of this study is to provide further insight into the correlates and predictors of young adults' eating habits, with particular emphasis on sociodemographics, reproductive health, and food upbringing.

ELIGIBILITY:
Inclusion Criteria:

* U.S. citizens
* Current, full-time, non-institutionalized residents of the United States
* Access to a computer with internet access

Exclusion Criteria:

* Non-U.S. citizens
* Non-resident of the United States
* No access to a computer with internet access

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The researchers aim to have the analyses be as nationally-representative as possible on certain criteria. To do so, there are goals for the number of participants belonging to 20 demographic profiles. The 20 demographic profiles will be based on sex assigned at birth (male, female), education (no college, some college +), and race/ethnicity (non-Hispanic white, non-Hispanic Black, non-Hispanic Asian, Hispanic, and non-Hispanic other). Using the 2019 American Community Survey, a nationally representative survey of adults in the United States, we have identified what proportion of 18- to 24-year-olds fall into each of the 20 demographic profiles. Taking these proportions, we will incorporate a 15% oversample of Black, Asian, and Hispanic individuals.
Sampling Method: Non-Probability Sample
Enrollment: 1123 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Diet quality | Baseline
  Diet quality as estimated using the Healthy Eating Index-2015, based on reported dietary intake.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hess, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT06096636/ICF_000.pdf